CLINICAL TRIAL: NCT03608098
Title: Long Pulse Versus Short Pulse Laser Dusting for Renal Stones
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Key study team members working on the study are leaving the institution.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Cogenix Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00049526
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2018-12

CONDITIONS: Kidney Stone; Ureter Stone; Renal Stone
Keywords: Basketing; Dusting; Holmium Laser; Laser Lithotripsy; Intracorporeal Lithotripsy; Urolithiasis
MeSH Terms: conditions — Kidney Calculi; Ureterolithiasis; Nephrolithiasis; Urolithiasis

STUDY DESIGN:
Intervention Model Description: All subjects enrolled in the study will be randomized to either short pulse or long pulse for treatment of their stones. The date of treatment will be decided between the subject and the treating surgeon. All treatments will be performed using the standard of care and will be performed in the same fashion as procedures for patients not enrolled in the study. There is no modification of the techniques used to remove the stones. Post operatively, we plan to discharge all subjects home from the recovery unit. All subjects will be seen one week to one month after surgery for stent removal and a low dose CT of the abdomen and pelvis to assess stone free rates which is standard for all stone patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Short Pulse Duration Group (Active Comparator): A short pulse duration (300 μs or 350 μs) will be used in this group.
  Interventions: Device: Short Pulse Duration
- Long Pulse Duration Group (Active Comparator): A long laser pulse duration (700 μs or 1500 μs) will be used in this group.
  Interventions: Device: Long Pulse Duration

INTERVENTIONS:
Device: Short Pulse Duration — The holmium laser device will be used on a short laser pulse duration setting (300 μs or 350 μs)
  Arms: Short Pulse Duration Group
Device: Long Pulse Duration — The holmuim laser device will be used on a long laser pulse duration setting (700 μs or 1500 μs)
  Arms: Long Pulse Duration Group

SUMMARY:
The purpose of this research study is to compare how well two treatments work for removing kidney stones. The two study groups include ureteroscopy with long/short pulse lithotripsy to remove kidney stones. Both of these options are considered standard of care and are used currently in surgery.

DETAILED DESCRIPTION:
This study will compare two types of laser lithotripsy to see the pulse duration to determine which settings are more effective. This is a randomized control trial with subjects randomized to either long pulse or a short pulse group. Those subjects with a single kidney/ureter stone measuring up to 20 mm will be eligible for the study. The procedures will be performed using the standard of care instruments and techniques but the pulse type setting in surgery will be constant. Some Holmium laser devices provide the option to modulate the pulse duration. A longer laser pulse duration (700 μs or 1500 μs) as compared to a traditional pulse duration (300 μs or 350 μs) has been demonstrated in vitro studies to provide effective stone disintegration while reducing laser fiber tip degradation and stone retropulsion. Both the long and the short setting can dust the stone and currently we alternate in each procedure from one setting to the other and it is unclear which setting is more effective. No changes to operative technique will be performed for subjects in the study vs regular patients undergoing the same procedure. All subjects will be seen one week to one month after surgery for stent removal and follow up.

ELIGIBILITY:
Inclusion Criteria:

* Kidney/ureter single stone between up to 2 cm
* Age over 18 years
* Two kidneys

Exclusion Criteria:

* Solitary Kidney
* Age under 18
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | 1 month after surgery
  Proportion of participants free of stones after procedure reported by group

SECONDARY OUTCOMES:
Operative duration time | 1 month after surgery
  Operative duration time measured by minutes
Need for Secondary Procedures | 1 month after surgery
  The number of participants needing additional secondary procedures will be reported per group

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gutierrez-Aceves, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson CP, Pace KT, Pais VM, Pearle MS, Preminger GM. American Urological Association (AUA) guideline surgical management of stones: American Urological Association Surgical Management 2016; April:1-50.
- [Background] Chew BH, Brotherhood HL, Sur RL, Wang AQ, Knudsen BE, Yong C, Marien T, Miller NL, Krambeck AE, Charchenko C, Humphreys MR. Natural History, Complications and Re-Intervention Rates of Asymptomatic Residual Stone Fragments after Ureteroscopy: a Report from the EDGE Research Consortium. J Urol. 2016 Apr;195(4 Pt 1):982-6. doi: 10.1016/j.juro.2015.11.009. Epub 2015 Nov 14. PMID 26585680
- [Background] Matlaga et al. Ureteroscopic Laser Lithotripsy: A Review of Dusting Versus Fragmentation With Extraction. Journal of Endourology. October 2017. Epub ahead of publication.
- [Background] Li R, Ruckle D, Keheila M, Maldonado J, Lightfoot M, Alsyouf M, Yeo A, Abourbih SR, Olgin G, Arenas JL, Baldwin DD. High-Frequency Dusting Versus Conventional Holmium Laser Lithotripsy for Intrarenal and Ureteral Calculi. J Endourol. 2017 Mar;31(3):272-277. doi: 10.1089/end.2016.0547. Epub 2017 Jan 16. PMID 27960541
- [Background] Wollin DA, Ackerman A, Yang C, Chen T, Simmons WN, Preminger GM, Lipkin ME. Variable Pulse Duration From a New Holmium:YAG Laser: The Effect on Stone Comminution, Fiber Tip Degradation, and Retropulsion in a Dusting Model. Urology. 2017 May;103:47-51. doi: 10.1016/j.urology.2017.01.007. Epub 2017 Jan 16. PMID 28089885